CLINICAL TRIAL: NCT02798276
Title: Efficacy of the Adipose Graft Transposition Procedure (AGTP) in Patients With a Myocardial Scar: The AGTP II Trial
Acronym: AGTP II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Antoni Bayés Genís (Other)
Responsible Party: Sponsor-Investigator, Antoni Bayés Genís, Antoni Bayes-Genis, Chief of the Cardiology Service, Germans Trias i Pujol Hospital
Organization: Germans Trias i Pujol Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ICOR-2016-01
Record Dates: First submitted 2016-05-26; First posted 2016-06-14 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; Cardiac regeneration; Cardiac surgery
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AGTP-treatment (Experimental): Patients in which the non-revascularizable area will be covered by the adipose graft and the revascularizable area will be treated with the normal procedure.
  Interventions: Procedure: AGTP-treatment
- Control (Other): Patients in with the non-revascularizable area will be left untouched and the revascularizable area will be treated normally.
  Interventions: Other: Control

INTERVENTIONS:
Procedure: AGTP-treatment — Patients with a myocardial necrosis candidates for revascularization of other myocardial areas, will be enrolled. The non-revascularizable area will be covered with the adipose graft and the revascularizable area will be treated with the normal procedure (by-pass).
  Arms: AGTP-treatment
Other: Control — Patients with a myocardial necrosis, candidates for revascularization of other myocardial areas, will be enrolled. The non-revascularizable area will be left untouched and the revascularizable area will be treated normally (by-pass).
  Arms: Control

SUMMARY:
The purpose of this trial is to evaluate the efficacy of a pericardial adipose graft transposition (Adipose Graft Trasposition Procedure, AGTP) for the improvement of cardiac function in patients with a chronic myocardial infarction. Preclinical studies in the porcine model of myocardial infarction have shown that the AGTP reduces infarct area and improves cardiac function. A first-in-man clinical (NCT01473433) trial showed that the AGTP is safe in patients.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age, capable of giving informed consent.
* Q wave in the ECG
* Myocardial infarct >=50% transmularity by NMR non revascularizable (for transmurality or bad vessel).
* Candidate to bypass for other myocardial areas

Exclusion Criteria:

* Severe non cardiac co-morbidity with a reduction of life expectancy of less than 1 year
* Severe valvular disease candidate for surgical restoration
* Candidate to ventricular remodeling
* Contraindication for NMR
* Severe renal or hepatic failure
* Abnoraml laboratory tests (no explanation at inclusion)
* Previous cardiac intervention
* Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Changes in necrotic mass ratio (%) by gadolinium retention. | 0-3-12 months
  necrotic mass ratio (%)

SECONDARY OUTCOMES:
Improvement in regional contractibility by NMR | 0-3-12 months
  regional contractibility
Changes in functional parameters by Nuclear Magnetic Resonance: ventricular ejection fraction | 0-3-12 months
  Left Ventricular Ejection Fraction, Right Ventricular Ejection Fraction (%)
Changes in functional parameters by Nuclear Magnetic Resonance: ventricular volumes | 0-3-12 months
  LVESV, LVEDV, RVESV, RVEDV (mL)
Changes in functional parameters by NMR: Cardiac output | 0-3-12 months
  L/min
Levels of natriuretic peptides | 0-1 week-3-12 months
  NTproBNP
Arrhythmia by 24-h Holter | 0--3-12 months
  Aupraventricular and ventricular arrhytmias
All-cause death or re-admission | 12 months
  All-cause death or >24h re-hospitalization due to all-cause
Cardiovascular death or re-admission | 12 months
  Cardiovascular death or >24h re-hospitalization due to cardiovascular causes

OTHER OUTCOMES:
Changes in infarct size: left ventricular necrotic mass | 0-3-12 months
  grams

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Germans Trias University Hospital; Germans Trias Research Institute, Badalona, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Son Espases Hospital, Palma de Mallorca
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid

REFERENCES:
- [Background] Bayes-Genis A, Galvez-Monton C, Prat-Vidal C, Soler-Botija C. Cardiac adipose tissue: a new frontier for cardiac regeneration? Int J Cardiol. 2013 Jul 15;167(1):22-5. doi: 10.1016/j.ijcard.2012.05.082. Epub 2012 Jun 17. PMID 22709728
- [Background] Galvez-Monton C, Prat-Vidal C, Roura S, Soler-Botija C, Llucia-Valldeperas A, Diaz-Guemes I, Sanchez-Margallo FM, Bayes-Genis A. Post-infarction scar coverage using a pericardial-derived vascular adipose flap. Pre-clinical results. Int J Cardiol. 2013 Jun 20;166(2):469-74. doi: 10.1016/j.ijcard.2011.11.019. Epub 2011 Dec 2. PMID 22137092
- [Background] Galvez-Monton C, Prat-Vidal C, Roura S, Farre J, Soler-Botija C, Llucia-Valldeperas A, Diaz-Guemes I, Sanchez-Margallo FM, Aris A, Bayes-Genis A. Transposition of a pericardial-derived vascular adipose flap for myocardial salvage after infarct. Cardiovasc Res. 2011 Sep 1;91(4):659-67. doi: 10.1093/cvr/cvr136. Epub 2011 May 16. PMID 21576133
- [Background] Bayes-Genis A, Gastelurrutia P, Camara ML, Teis A, Lupon J, Llibre C, Zamora E, Alomar X, Ruyra X, Roura S, Revilla A, San Roman JA, Galvez-Monton C. First-in-man Safety and Efficacy of the Adipose Graft Transposition Procedure (AGTP) in Patients With a Myocardial Scar. EBioMedicine. 2016 May;7:248-54. doi: 10.1016/j.ebiom.2016.03.027. Epub 2016 Apr 10. PMID 27322478
- [Background] Ma H, Liu J, Qian L. Fat for fostering: Regenerating injured heart using local adipose tissue. EBioMedicine. 2016 May;7:25-6. doi: 10.1016/j.ebiom.2016.03.024. Epub 2016 Mar 20. No abstract available. PMID 27322455
- [Derived] Gastelurrutia P, Galvez-Monton C, Camara ML, Bustamante-Munguira J, Garcia-Pavia P, Avanzas P, Alberto San Roman J, Pascual-Figal D, Teresa E, Crespo-Leiro MG, Manito N, Nunez J, Fernandez-Aviles F, Caballero A, Teis A, Lupon J, Brugada R, Martin C, Silva J, Revilla-Orodea A, Canovas SJ, Melero JM, Cuenca-Castillo JJ, Gonzalez-Pinto A, Bayes-Genis A. Rationale and design of a multicentre, prospective, randomised, controlled clinical trial to evaluate the efficacy of the adipose graft transposition procedure in patients with a myocardial scar: the AGTP II trial. BMJ Open. 2017 Aug 4;7(8):e017187. doi: 10.1136/bmjopen-2017-017187. PMID 28780562